CLINICAL TRIAL: NCT04015414
Title: Varenicline Versus Cytisine for Smoking Cessation in the Primary Care Setting in Croatia and Slovenia - a Randomized Controlled Trial
Brief Title: Varenicline Versus Cytisine for Smoking Cessation in Primary Care Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other); University of Zagreb School of Medicine (Unknown); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Stjepan Oreskovic, Full Professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRAND / MEF Zagreb - LPPHR2018; WI231434 IIR (Other Grant/Funding Number: Pfizer Inc., a Delaware corporation with an office of business at 235 East 42nd Street, New York, NY 10017 ("Pfizer")
Record Dates: First submitted 2019-07-02; First posted 2019-07-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; cytisine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Varenicline (Champix) (Active Comparator): Varenicline treatment will start one week prior to the patient's target quit date at 0.5 mg/day for days 1-3, 0.5 mg twice daily for days 4-7. On the target quit date (day 8), the dose will be increased to 1 mg twice daily and maintained for day 8-week 12. Patients will receive weekly calls during the first 4 weeks and at weeks 8, 12, and 24 to inquire about medication adherence and smoking status, motivate the patient to take the medication, encourage them not to smoke, and ask about possible side effects or other issues.
  Interventions: Drug: Varenicline
- Cytisine (Tabex) (Active Comparator): Patients will be asked to reduce their smoking during the first 4 days of treatment with aim to quit on the 5th day (target quit date). Cytisine treatment will follow standard manufacturer's dosing protocol of one tablet every 2 hours through the waking day (up to 6 tablets per day) for days 1-3, one tablet every 2.5 hours (up to 5 tablets per day) for days 4-12, one tablet every 3 hours (up to 4 tablets per day) for days 13-16, one tablet every 4-5 hours (3 tablets per day) for days 17-20, and one tablet every 6 hours (2 tablets per day) for days 21-25.
  Interventions: Drug: Cytisine

INTERVENTIONS:
Drug: Varenicline — 191 patients will receive varenicline for 12 weeks and regular phone calls with brief counseling Tabex: 188 patients will receive cytisine for 25 days and regular phone calls with brief counseling
  Other Names: Champix
  Arms: Varenicline (Champix)
Drug: Cytisine — 185 patients will receive cytisine for 25 days and regular phone calls with brief counseling
  Other Names: Tabex
  Arms: Cytisine (Tabex)

SUMMARY:
The overall goals of this study are to 1) assess awareness of interest in the use of pharmacotherapy for smoking cessation in Croatia and Slovenia, countries in Central Europe with very high smoking prevalence, and 2) investigate whether cytisine is at least as feasible and effective as varenicline in helping smokers to quit in a real-life setting: family medicine practices in Croatia and Slovenia. The investigators propose to survey patients from 40 primary care practices (20 in Croatia and 20 in Slovenia) to assess desire to quit smoking and awareness and interest in pharmacotherapy. Additionally, 380 patients with interest in quitting smoking will be randomly assigned to use varenicline or cytisine to help quit smoking.

The investigators hypothesize that cytisine is at least as feasible and effective as varenicline in helping smokers from primary care practices in Croatia and Slovenia to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Receive care in one of forty family medicine practices in Croatia and Slovenia
* Aged 18 or older
* Current smokers
* Indicate a desire to stop smoking and to use pharmacotherapy.

Exclusion Criteria:

* Mental illness who cannot provide informed consent for the study
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Seven day abstinence from tobacco | 12-weeks following target quit date
  Proportion of patients in the varenicline and cytisine groups who self-report seven-day abstinence from tobacco.

SECONDARY OUTCOMES:
Seven day abstinence from tobacco country and practice | 4-weeks following target quit date
  Proportion of patients in the varenicline and cytisine groups who self-report seven-day abstinence from tobacco.
Seven day abstinence from tobacco | 8-weeks following target quit date
  Proportion of patients in the varenicline and cytisine groups who self-report seven-day abstinence from tobacco.
Seven day abstinence from tobacco | 24-weeks following target quit date
  Proportion of patients in the varenicline and cytisine groups who self-report seven-day abstinence from tobacco.
Seven day abstinence from tobacco | 4, 8, 12, and 24 weeks following target quit date
  Repeated measures of proportion of patients in the varenicline and cytisine groups who self-report seven-day abstinence from tobacco
Continuous smoking cessation | 4, 8, 12, and 24 weeks following target quit date
  Proportion of patients who self-report continuous smoking cessation in the varenicline and cytisine groups (5 cigarettes allowed)
Medication adherence | 1, 2, 3, 4, 8, 12 weeks following target quit date
  Self report of adherence to assigned treatment protocol, including count of pills and stopping treatment (including reasons)
Side effects | 4, 8, 12, and 24 weeks following target quit date
  Self-report of any unintended sign, symptom, or other health-related issue that occurs during treatment with varenicline or cytisine

CONTACTS AND LOCATIONS:
Overall Officials: Stjepan Oreskovic, PhD, Principal Investigator — University of Zagreb School of Medicine; Sanja Percac Lima, PhD, MD, Principal Investigator — Massachusetts General Hospital; Hrvoje Tiljak, PhD, Study Chair — University of Zagreb School of Medicine; Janez Rifel, PhD, Study Chair — University of Ljubljana School of Medicine; Jeffrey M Ashbruner, PhD, MPH, Study Chair — Massachusetts General Hospital; Zalika Klemenc Ketis, MD, PhD, Study Chair — University of Ljubljana School of Medicine; Tin Oreskovic, Study Chair — IBM Chief Analytics Office, MIT-IBM AI Lab
Locations (2):
- University of Zagreb School of Medicine, Zagreb, Croatia
- University of Ljubljana School of Medicine, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the data collection and analysis